CLINICAL TRIAL: NCT05603494
Title: The Use of Home Spirometry in the Monitoring of Patients With Acute Exacerbation of Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202200852B0
Record Dates: First submitted 2022-08-02; First posted 2022-11-02 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Asthma Attack

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- home spirometry group (Experimental)
  Interventions: Device: NuvoAir

INTERVENTIONS:
Device: NuvoAir — Use of NuvoAir in pulmonary function monitoring during asthma attack

SUMMARY:
After outpatient clinic visit, asthmatic patients with worsening of symptoms (including dyspnea, wheezing, chest tightness, cough, activity limitation, awaken in the midnight due to discomfort) and are diagnosed of acute exacerbation by physician, will be recruited. The patients are asked to record symptoms using asthma symptom diary (ASD) with home spirometry simultaneously for 14 days.

Visit 1 (day 1)

All patients will be evaluated the following:

1. Record the patients' demographics (age, gender, race), baseline characteristics, comorbidities, health care resources use (visits, lab tests, hospitalization and cost), pharmacological and non-pharmacological treatments
2. Blood sampling for eosinophils, eosinophil cationic protein (ECP) and immunoglobulin E (IgE) as clinically indicated (if no data available within one year for the last two)
3. The study assistant will introduce to the patient how to manipulate the home spirometry and its app, and to record the daily asthma symptoms by using the ASD on the mobile phone.

Visit 2 (day 15) All patients will be arranged outpatient clinic follow up 2 weeks later from the first visit. The outpatient clinic physician will check the home spirometry report and ASD symptom score in the past 2 weeks, and have a well explanation of these results.

Statistical analysis The usage of digital function including input ASD, and the lung function from portable spirometer in study arm will be demonstrated by descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 75 years old asthmatic patients under regular treatment for at least 3 months.
* Patients in asthma acute exacerbation (symptoms onset within 1 week) and received oral corticosteroid for more than 3 days.

Exclusion Criteria:

* Refuse to provide inform consent.
* Patients with chronic obstructive pulmonary disease.
* Patients who receive more than 20mg prednisone or equivalent dose per day.
* Patients who are incapable of using smart phone.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
To compare between changes in asthma symptoms and pulmonary function by home spirometry | 2 weeks
  To compare between changes in asthma symptoms by asthma symptom diary (scoring in points) and changes in forced expiratory volume in 1 second (FEV1, in liters) in patients with acute exacerbation of asthma.
  Asthma symptom diary (ASD) consist of daytime and nighttime score will be recorded everyday over the 14-day study period.

SECONDARY OUTCOMES:
To compare the changes in daily asthma rescue medication use and pulmonary function by home spirometry | 2 weeks
  To compare between changes in the daily inhalation times (puffs in times per day) and changes in forced expiratory volume in 1 second (FEV1, in liters) in patients with acute exacerbation of asthma.
  Rescue medication (Fenoterol, Albuterol, inhaled corticosteroid-formoterol) use was measured by the number of inhalations per day.

OTHER OUTCOMES:
To compare the degree of discrepancy between different asthma phenotypes | 2 weeks
  To compare between changes in asthma symptoms (scoring in points) and forced expiratory volume in 1 second (FEV1, in liters) in patients with acute exacerbation of asthma in different asthma phenotypes (allergic type, non-allergic T2 type, non-T2 type).

CONTACTS AND LOCATIONS:
Locations (1):
- Chiung-Hung, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Brouwer AF, Roorda RJ, Brand PL. Home spirometry and asthma severity in children. Eur Respir J. 2006 Dec;28(6):1131-7. doi: 10.1183/09031936.06.00118205. Epub 2006 Jul 26. PMID 16870659
- [Result] Park SY, Yoon SY, Shin B, Kwon HS, Kim TB, Moon HB, Cho YS. Clinical factors affecting discrepant correlation between asthma control test score and pulmonary function. Allergy Asthma Immunol Res. 2015 Jan;7(1):83-7. doi: 10.4168/aair.2015.7.1.83. Epub 2014 Nov 25. PMID 25553267